CLINICAL TRIAL: NCT05019547
Title: Validity and Reliability of the Turkish Version of the Inflammatory Arthritis Facilitators and Barriers to Physical Activity
Brief Title: The Turkish Version of the Inflammatory Arthritis Facilitators and Barriers to Physical Activity
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK 2021 - 15
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Axial Spondyloarthritis: Participants with Axial Spondyloarthritis
  Interventions: Behavioral: Determining Barriers and Facilitators of Physical Activity

INTERVENTIONS:
Behavioral: Determining Barriers and Facilitators of Physical Activity — Determining Barriers and Facilitators of Physical Activity

SUMMARY:
Our aim in this study is to translate the Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) Questionnaire which was developed to determine the factors that facilitate and prevent individuals for physical activity for patients with inflammatory arthritis into Turkish language. Also, our aim is to evaluate the validity and reliability of the IFAB Questionnaire in the Turkish population, and to perform a cultural adaptation if necessary at the same time. Determining the factors that facilitate and prevent individuals for physical activity interventions with rheumatic diseases and then designing physical activity programs considering these factors may play an important role in reducing the symptoms caused by the disease and increasing their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Diagnosed with Axial Spondyloarthritis by an experienced rheumatologist
* To have the neurological competence and cognitive level to answer the scale questions.

Exclusion Criteria:

* Having a rheumatological disease other than Axial Spondyloarthritis ,
* Using an assistive device for walking.
* Any verbal or written communication problems in Turkish,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Axial Spondyloarthritis
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory Arthritis Barriers and Facilitators to Physical Activity Questionnaire (IFAB) | 1 day
  The IFAB Questionnaire was developed by Davergne et al. in 2020 and aims to evaluate the factors that facilitate or prevent physical activity in individuals with inflammatory arthritis. The IFAB questionnaire consists of 10 items. Of these 10 items, 4 were identified as potential barriers or facilitators, 3 as only barriers and 3 as only facilitators. The participant is asked to rate how much the item facilitates or prevents from physical activity between 0 and 10, "0" has no effect on physical activity, and "10" has maximum (negative or positive) effect on physical activity. A high score from the questionnaire indicates that the facilitators are at a high level and the barriers are at a low level.
The Exercise Benefits or Barriers Scale | 1 day
  The Exercise Benefits and Barriers Scale has been developed by Sechrist et al. and the Turkish validity and reliability studies were conducted by Ortabağ et al. This scale will be used to evaluate criterion validity which evaluates the benefits and barriers of exercise perceived by the individual on a 4-point Likert-type scale with 43 questions. Scoring is performed as barrier score, benefit score and total score. A low score means less perceived barriers to exercise and greater benefits.
International Physical Activity Questionnaire - Short Form | 1 day
  The physical activity level reported by the participants will be evaluated with the International Physical Activity Questionnaire - Short Form. The International Physical Activity Questionnaire - Short Form questions the time spent walking, moderate and vigorous activities, and sitting with 7 questions. The duration (minutes) and frequency (days) of each activity are questioned. The physical activity levels of the participants will be classified as inactive, minimally active and very active according to the results.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 1 day
  The HADS scale was developed to assess anxiety and depression in individuals without psychiatric illness. Of the 14-item questionnaire, 7 questions assess depression and 7 questions assess anxiety and each response consists of a four-point rating scale (0 to 3); a higher score indicates a worse condition.For each subscale the total score is at most 21.
Health Assessment Questionnaire - Disability Index | 1 day
  This questionnaire evaluates the level of functional disability in patients with rheumatological disease over 20 questions. It determines the level of difficulty of the person during the activities that are most frequently performed in daily life such as dressing, eating, hygiene, walking, sitting up, reaching and grasping. A high score indicates a low level of functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk O, Feyzioglu O, Saritas F. Inflammatory Arthritis Facilitators and Barriers (IFAB) for physical activity questionnaire: cross-cultural adaptation into Turkish and evaluation of its psychometric properties. Disabil Rehabil. 2023 Aug;45(17):2818-2825. doi: 10.1080/09638288.2022.2104940. Epub 2022 Aug 1. PMID 35914576